CLINICAL TRIAL: NCT07289659
Title: Arthroscopic Repair of Partial Thickness Articular Side Rotator Cuff Tears Using Transtendon Versus Conversion Repair Techniques.
Brief Title: Arthroscopic Repair of Partial Thickness Articular-Side Rotator Cuff Tears: Transtendon Versus Conversion Repair Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Ahmed El-Desouky, Associate Professor of Orthopedic surgery, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N-383-2019
Record Dates: First submitted 2025-11-15; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Partial Thickness Articular-Side Rotator Cuff Tears

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conversion Repair (Active Comparator): Patients with PT-RCTs treated using the arthroscopic conversion technique.
  Interventions: Procedure: Arthroscopic Conversion Repair
- Transtendon Repair (Active Comparator): Patients with PT-RCTs treated using the arthroscopic transtendon repair technique.
  Interventions: Procedure: Arthroscopic Transtendon Repair

INTERVENTIONS:
Procedure: Arthroscopic Conversion Repair — Patients undergo arthroscopic conversion repair, where the partial-thickness tear is converted to a full-thickness tear and repaired using standard arthroscopic techniques.
  Arms: Conversion Repair
Procedure: Arthroscopic Transtendon Repair — Patients undergo arthroscopic transtendon repair, preserving the intact bursal surface of the tendon while repairing the articular-side defect using suture anchors.
  Arms: Transtendon Repair

SUMMARY:
This prospective randomized clinical trial compared two arthroscopic techniques for repairing partial-thickness articular-side rotator cuff tears: transtendon repair and conversion repair. Eligible patients with symptomatic tears exceeding 50% of tendon thickness, confirmed by MRI and intraoperative assessment, were randomly assigned to either repair technique. Functional outcomes, range of motion, complications, and MRI healing were assessed up to 24 months postoperatively

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering symptomatic PT-RCTs exceeding 50% of the tendon thickness, documented by preoperative magnetic resonance imaging (MRI) and confirmed by arthroscopy intraoperative.
* Failure of nonoperative management for at least 3 months.

Exclusion Criteria:

* Prior shoulder surgery.
* Severe concomitant pathologies including glenohumeral arthritis, advanced subscapularis tear, and biceps tendon rupture.
* Associated Bankart lesion.
* Patients with uncontrolled Diabetes mellites.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeons (ASES) Score | Baseline and 24 months postoperatively
Constant-Murley Score (CMS) | Baseline and 24 months postoperatively
Visual Analogue Scale (VAS) for Pain | Baseline and 24 months postoperatively

SECONDARY OUTCOMES:
Range of Motion (ROM) | Preoperative and 24 months postoperatively.
  Measure the range of:
  1. Forward flexion
  2. Abduction
  3. External rotation
  4. Internal rotation
Complication Rate | Up to 24 months postoperatively
  Number of cases with:
  Stiffness Persistent pain Infection
MRI Healing Status | 12 months postoperatively
  Number of cases with complete healing in MRI

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Alainy, Cairo, Egypt